CLINICAL TRIAL: NCT04095845
Title: A Prospective Randomised Controlled Trial Comparing Computerised Tomography Based Planning of Conventional Total Hip Arthroplasty Versus Mako Robotic-arm Assisted Total Hip Arthroplasty
Brief Title: Conventional Total Hip Arthroplasty vs Mako Robotic-arm Assisted Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Stryker Instruments (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17/0766
Record Dates: First submitted 2019-07-17; First posted 2019-09-19 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis, Hip; Osteoarthritis; Surgery
Keywords: total hip arthroplasty; total hip replacement; implant position; computerised tomography; makoplasty; robotic surgery
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CO THA (Active Comparator): Computerised tomography based planning of conventional total hip arthroplasty
  Interventions: Device: CO THA
- Mako THA (Experimental): Mako robotic-arm assisted total hip arthroplasty
  Interventions: Device: Mako THA

INTERVENTIONS:
Device: CO THA — Replacement of arthritic hip with artificial implant using CT-based navigation and conventional technique
  Arms: CO THA
Device: Mako THA — Replacement of arthritic hip with artificial implant using mako robotic-arm assist
  Arms: Mako THA

SUMMARY:
The overall aim of this single-centre, prospective randomised controlled trial is to compare clinical, functional, and radiological outcomes in CO THA versus Mako THA. Patients undergoing Mako THA will form the investigation group and those undergoing CO THA will form the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patient has hip osteoarthritis requiring primary THA

  * Patient and surgeon are in agreement that THA is the most appropriate treatment
  * Patient is fit for surgical intervention following review by surgeon and anaesthetist
  * Patient age: Patients 18-80 years of age inclusive
  * Gender: male and female
  * Patient must be capable of giving informed consent and agree to comply with the postoperative review program
  * Patient must be a permanent resident in an area accessible to the study site
  * Patient must have sufficient postoperative mobility to attend follow-up clinics and allow for radiographs to be taken

Exclusion Criteria:

* Patient is not suitable for primary THA e.g. patient requires revision surgery for previously failed THA

  * Patient is not medically fit for surgical intervention
  * Patients under the age of 18 or over 80 years of age
  * Patient is immobile or has another neurological condition affecting musculoskeletal function
  * Patient is already enrolled on another concurrent clinical trial
  * Patient is unable or unwilling to sign the informed consent form specific to this study
  * Patient lacks capacity to give informed consent
  * Patient is unable to attend the follow-up programme
  * Patient is non-resident in local area or expected to leave the catchment area postoperatively

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Reproducibility of the planned pre-operative centre of rotation [COR] of the hip | 6 weeks post-op
  Radiographic assessment of the COR will be performed using coronal plane images from the preoperative pelvic CT scan and postoperative CT scanogram at six weeks after surgery.
  The COR will be determined using the centre of a circle encompassing the native femoral head on the contralateral side in the preoperative films and the prosthetic femoral head on the ipsilateral side on postoperative films. The horizontal COR will be calculated by measuring the distance between the COR and a line running directly perpendicular from the midline of the pelvis, which is defined as a line connecting the middle of the pubic symphysis and the middle of the inter-sacroiliac line. The vertical COR will be calculated by measuring the distance of a line that runs directly perpendicular from the inter-tear drop line to the COR.

SECONDARY OUTCOMES:
Spinopelvic alignment | Preoperatively and postoperatively at 6 months
  Spinopelvic alignment with plain radiographs in sitting and standing position;
  1. standing anteroposterior [A/P] lumbar spine and pelvis
  2. standing lateral lumbar spine and pelvis
  3. seated lateral lumbar spine and pelvis
Operating time | Intraoperative
  Length of operating time in minutes
Blood loss | Intraoperative
  Estimated intraoperative blood loss in millilitres [ml]
Blood transfusion requirements | Intraoperative
  Units of blood required for transfusion intraoperatively; in whole units
Bone resection thickness | Intraoperative
  Thickness of bone resected during the surgical procedure in millimetres
Length of hospital stay | 6 weeks post op
  Length of patient hospital stay from admission to documented discharge; hours
Oxford hip score [OHS] | Pre-op; 6 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Patient recorded outcome measure via questionnaire. Scored 0-48 with 0 = poor score and 48 = best possible score
Harris Hip Score [HHS] | Pre-op; 6 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Patient recorded outcome measure via questionnaire. Scored 0-100 with 100 best possible outcome
Western Ontario and Mcmaster Universities Osteoarthritis Index [WOMAC] | Pre-op; 6 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Patient recorded outcome measure via questionnaire. Questions regarding pain, stiffness and disability of affected hip joint. 0= best possible score
University of California at Los Angeles hip [UCLA] | Pre-op; 6 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Patient recorded outcome measure via questionnaire. Score 0-10 with 10 being best possible outcome, 0 being worst possible outcome
European Quality of Life questionnaire with 5 dimensions for adults [EQ-5D] | Pre-op; 6 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Health-related quality of life patient recorded outcome measure via questionnaire. Score 0-1 with 1 being best possible outcome and 0 being worst possible outcome
Complications | Intraoperative; 6 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Complications relating to surgery; to include development of:
  leg-length inequality in millimetres; deep venous thrombosis; fracture; dislocation of the prosthesis; neurovascular injury; infection of wound; deep infection involving prosthesis; re-operation or revision surgery; pulmonary embolus; heart attack; stroke; death

CONTACTS AND LOCATIONS:
Overall Officials: Fares S Haddad, Study Chair — UCL Hospital NHS Foundation Trust; Babar Kayani, Principal Investigator — UCL Hospitals NHS Foundation TRust
Locations (1):
- UCL Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD

REFERENCES:
- [Derived] Kayani B, Konan S, Tahmassebi J, Ayuob A, Haddad FS. Computerised tomography-based planning with conventional total hip arthroplasty versus robotic-arm assisted total hip arthroplasty: study protocol for a prospective randomised controlled trial. Trials. 2020 Sep 10;21(1):776. doi: 10.1186/s13063-020-04702-7. PMID 32912292